CLINICAL TRIAL: NCT05207501
Title: Intermittent Hypoxic vs Blood Flow Restriction vs Eccentric Moderate-intensity Exercise in Elderly
Brief Title: Effects of Different Moderate-intensity Exercise Methods on Health in the Elderly
Acronym: 4MIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Gregoire Millet, Associate Professor, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-02135
Record Dates: First submitted 2021-12-23; First posted 2022-01-26 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Healthy Aging
Keywords: Hypoxia; Blood Flow Restriction; Eccentric cycling; Exercice; Elderly
MeSH Terms: conditions — Hypoxia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized parallel group active-control study.
Who Masked: Participant
Masking Description: The active-control group will receives a comparable standard treatment to the three other groups: Moderate Intensity Interval Training on a ergocycle without any additional feature.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate-intensity intermittent training (MIIT) (Active Comparator): The MIIT will be conducted on a cycle ergometer (Lode Ex. calibur Sport Ergometer, Lode B.V., the Netherlands) in normoxia (FiO2 = ~ 21%). The participants will perform the MIIT starting with the ergometer resistance set to obtain the %HRmax set (~75-80%) during 5 minutes and will rest 5 minutes after each interval of exercise. The HRmax will be considered as 200 - age.
  Interventions: Behavioral: Exercise
- MIIT during intermittent hypoxic exposure (IHYP + MIIT) (Experimental): A normobaric hypoxic chamber (ATS Altitude Training, Sydney, Australia) will be used for this protocol. The chamber (2.4 m x 5 m x 2.5 m) allows, via a filter and compressor system, to extract oxygen molecules and to reduce the fraction of inspired oxygen (FiO2) with no modification of the barometric pressure.
  Interventions: Behavioral: Exercise
- MIIT during intermittent blood flow restriction (IBFR + MIIT) (Experimental): The IBFR + MIIT protocol will be performed while cycling in normoxia (FiO2 = ~ 21%). Elastic, pneumatic cuffs (BStrong, Park City, Utah, USA) will be administered as high as possible at the inguinal crease of the upper thigh and will be inflated during the cycling to the set pressure of 400 mmHg (except for the first training session, it will be of 250 mmHg to minimize soreness and to accustom patients to vascular occlusion training). The cuffs will be deflated at interval rest.
  Interventions: Behavioral: Exercise
- Moderate-intensity eccentric cycling (MIEC) (Experimental): The MIEC will be conducted on a cycle ergometer (Excalibur, Lode, Groningen, The Nederlands) in normoxia (FiO2 = ~ 21%). The participants will be instructed to resist against the pedal movement (cadence set at 15 revolutions/min) to produce the required torque (set to obtain the 75-80%HRmax) indicated by visual feedback for 5 minutes and will rest 5 minutes after each interval of exercise. The HRmax will be considered as 200 - age. The HR responses will be monitored (Polar Electro Oy, Kempele, Finland).
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will perform 3 times a week for 4 weeks a moderate intensity interval training.

SUMMARY:
Aging is linked to a higher risk of cardiovascular disease. Physical exercise is recognized as an excellent strategy to prevent cardiovascular diseases and cognitive aspects, generating healthier elderly people. The beneficial effects of physical training seem to be greater when performed:

* In hypoxic conditions (i.e. when the amount of oxygen in the air is decreased as at altitude).
* With intermittent blood flow restriction (by inflating pneumatic cuffs around the thighs to a pressure that restricts blood flow). This equipment is harmless.
* With eccentric training (resisting against the movement of the pedal of a bicycle rather than pushing it).

The purpose of this study is then to evaluate whether moderate intensity intermittent training can induce similar or greater effects on cardiovascular health when combined with intermittent hypoxia, intermittent blood flow restriction or eccentric training.

DETAILED DESCRIPTION:
Aging is associated with a higher risk of cardiovascular disease due mainly to high blood pressure. Physical exercise is recognized as an excellent non-pharmacological strategy to prevent cardiovascular disease and cognitive aspects, thus generating healthier elderly people.

* Interestingly, living at altitude seems to reduce some cardiovascular risks. In addition, the beneficial effects of physical training seem to be greater when performed under hypoxic conditions (i.e. when the amount of oxygen in the air is decreased as at altitude).
* Another interesting strategy for the elderly is intermittent blood flow restriction. This involves inflating pneumatic cuffs around the limb(s) to a pressure that blocks or restricts blood flow to the affected muscles, alternating with rest phases. It has been found that endurance training, combined with blood flow restriction, promotes the growth of new blood vessels, which could be particularly important for the prevention of cardiovascular disease in the elderly, which is unfortunately common.
* Eccentric training is currently emerging as a promising training strategy for the elderly. It consists of resisting the movement of the pedal of a bicycle rather than pushing it. It requires less energy effort than traditional exercise with the same workload. Eccentric training has been shown to improve older adults' body composition and muscle strength, thereby improving exercise capacity and quality of life.

These training strategies may be of interest for cardiovascular health in older adults. However, there are few data on their combined effects with exercise in the elderly and there is no consensus to favor one method over another.

The objective of this study is then to evaluate whether moderate-intensity intermittent training can induce similar or superior effects on health indicators when combined with intermittent hypoxia, partial vascular occlusion, or eccentric training.

ELIGIBILITY:
Inclusion Criteria:

1. to be aged between 65 and 75 years old
2. not involved in regular physical activities for at least 6 months (i.e., doing no physical exercise over twice per week);
3. free of injuries as well as cardiovascular and respiratory disorders or central nervous system disease or receiving β-blocker medication;
4. not using dietary supplements, smoking or drugs which interfere with the measurements;
5. not using creatine supplementation, anabolic steroids, drugs, or medication with potential effects on physical performance;
6. to have body index mass between 20 and 30 kg/m²;
7. not to live above 800m of altitude;
8. to be vaccinated against COVID-19 and to have no symptoms (fever, cough, fatigue, loss of smell or taste);
9. able to complete all sessions;
10. able to give consent.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure [mmHg] | 4 weeks
  a major risk factor, when too high, for cardiovascular diseases.
Baroreflex sensitivity | 4 weeks
  A measurement of the mechanism that regulates acute blood pressure changes linked to the development and progression of cardiovascular diseases
Flow-mediated dilation | 4 weeks
  RHI index: a measure for arterial endothelial function
Heart rate variability | 4 weeks
  An independent predictor of cardiovascular mortality and sudden cardiac death.
6-Minute Cycle Test [km] | 4 weeks
  an estimation of the maximal aerobic capacity
Knee flexion and extension isokinetic strength [N] | 4 weeks
  The knee flexion and extension strength will be measured with an isokinetic dynamometer
Muscle mass [kg] | 4 weeks
  An analysis of muscle mass will be done using DXA scan
Body fat [kg] | 4 weeks
  An analysis of body fat will be done using DXA scan

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No